CLINICAL TRIAL: NCT04566198
Title: Smoking in the Paris Fire Brigade and Comparison According to the Type of Service (Permanent or On-call)
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PPRC12; 2020-A01843-36 (Other: IDRCB)
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — The participants will have to filled out a questionnaire about their working conditions and their lifestyle habits.

SUMMARY:
Tobacco use is one of the world's leading preventable causes of disease and premature death, and the physician has a central role in detecting smokers and helping them to quit.

Tobacco use in the military undermines fitness, readiness and performance, and increases health care costs.

A study conducted on a French Army contingent on external operations in Afghanistan have shown an increase in tobacco use in situation of operational constraints (stress, shift work, etc.). However, another study conducted in Ivory Coast on a mobile gendarmerie squadron showed no significant difference.

Among the American firefighters who have been exposed to the 9/11 World Trade Center attacks, smoking have been shown to play an aggravating role in the recovery of lung function.

This study is aimed at assessing smoking prevalence in the Paris Fire Brigade, which is composed of young and healthy sportsmen and women who are exposed to strong operational constraints.

ELIGIBILITY:
Inclusion Criteria:

* To be 18 years of age or older
* To be French
* To be an active military member
* To work in the Paris Fire Brigade

Exclusion Criteria:

* To be a civilian
* To be a reservist
* To be a foreigner

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of active military members of the Paris Fire Brigade.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Proportion of smokers | At enrollment (day 1)
  The smoking status (smoker or non-smoker) will be determined according to the responses to the questionnaire. The proportion of smokers will be calculated by dividing the number of smokers by the total number of participants.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Médical de Champerret, Paris
  - Antenne médicale de Ménilmontant, Paris

IPD SHARING:
Plan to Share IPD: Undecided